CLINICAL TRIAL: NCT02821637
Title: Impact of an Effort Rehabilitation Program for Overweight or Obese Children and Teens on Quality of Life and Wellbeing: A French Monocentric Prospective Study
Brief Title: Impact of an Effort Rehabilitation Program for Overweight/Obese Children/Teens on Quality of Life and Wellbeing
Acronym: PRESEVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHRMSA 754; 2014-A01695-42 (Other: France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2016-06-20; First posted 2016-07-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2017-07

CONDITIONS: Pediatric Obesity
Keywords: teens; effort rehabilitation; quality of life; wellbeing; physical skills assessment
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Effort rehabilitation program (Other): An effort rehabilitation program designed for obese and overweight children or teens : 13 weekly sessions of 1hour30 then 1 session 2 months, 6 months and 12 months later.
  This program is part of the routine practice of the Pediatric Obesity and Pediatric Diabetes Organization of Mulhouse.
  Child Health Questionnaire (CHQ) of quality of life are completed by parents and children on the 1st and the 13th session, then 3 more times : 2, 6 and 12 months after the 13th session.
  Eurofit tests of Physical Fitness performed on the 1st and the 13th session, then 3 more times : 2, 6 and 12 months after the 13th session.
  Interventions: Other: Eurofit Tests of Physical Fitness (Eurofit); Behavioral: Child Health Questionnaire (CHQ); Other: Effort rehabilitation program

INTERVENTIONS:
Other: Eurofit Tests of Physical Fitness (Eurofit) — Eurofit tests are a physical skills assessment. For the study, tests performed on the 1st and the 13th session of the program, then 3 more times : 2 months, 6 months and 12 months after the 13th weekly session.
Behavioral: Child Health Questionnaire (CHQ) — The CHQ is a questionnaire about quality of life. The CHQ children form (CHQ-CF87) and the CHQ parent form (CHQ-PF50) are completed each time the Eurofit tests are performed : at the 1st and 13th weekly session then 2 months, 6 months and 12 months later.
Other: Effort rehabilitation program — Part of the routine practice of the Pediatric Obesity and Pediatric Diabetes Organization of Mulhouse, the program consists in 13 sessions of 1hour30 of adapted physical activity. The physical activity in this program use cycles of games where rules are adapted to the overweight or obese children. The activities are performed in a playful atmosphere, for example using creative games like tchoukball or peteca, with each session aiming a specific objective each time.

SUMMARY:
Obese and overweight children or teens can join the Prevention and Care of Pediatric Obesity and Pediatric Diabetes Organization of Mulhouse. Those patients who are no longer able to exercize because of their physical condition start an effort rehabilitation program at the Organization. The study will evaluate the impact of this rehabilitation program on quality of life and appetency to physical activity for these children and teens.

DETAILED DESCRIPTION:
Because of a National Obesity Plan (2010-2013) initiated by the French government in charge of health, the Pediatric Obesity and Pediatric Diabetes Organization of Mulhouse was created in 2011.

This Organization is in charge of children or teens with:

* severe or growing obesity associated with respiratory, osteo-articular metabolic complications
* comorbidities worsened by obesity

The Organization and the Physical Medicine and Rehabilitation department of the Mulhouse Hospital have worked together to create an effort rehabilitation program for obese or overweight children. The program, aiming movement rehabilitation, is based on reinforcement and endurance activities in a playful atmosphere and in an important motivational dimension. A medical examination is performed before the first session to confirm the patient's ability to follow an effort rehabilitation program. Each session is supervised by a teacher of adapted physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 97 percentile
* at least one of the following symptoms :

  * respiratory functional signs
  * orthopedic complications
  * sleep apnea
  * cardiovascular complications
  * metabolic syndrome

Exclusion Criteria:

* lack of motivation
* uncontrolled psychological issue
* ambulatory care more appropriate to treat the same issues
* any related psychiatric pathology likely to worsen with weight loss
* patient or family not committed to therapeutics program
* psychological inability to deal with separation
* behavior disorders making collective activity impossible

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Evolution in the score of the Child Health Questionnaire (CHQ) of quality of life | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Appetency to physical activity assessed with the evolution of the amount of time spent weekly in a physical activity | Through study completion, an average of 1 year
Aerobic and physical capacities assessed with the Eurofit tests results | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study results — https://ecrin.app.unistra.fr/search/notice/view/ecrin-ori-343907